CLINICAL TRIAL: NCT05434143
Title: Chorus Sleep Randomized Controlled Trial
Brief Title: Chorus Sleep Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chorus Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-0001
Record Dates: First submitted 2022-05-11; First posted 2022-06-27 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sleep Disturbance
Keywords: mindfulness; breathwork; meditation
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Masking Description: This is a waitlist controlled design to a behavioral intervention. Assignment will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chorus Sleep (Experimental): During the 6-week intervention, participants will receive daily reminders to complete their daily sleep log and a link to a chorus sleep class for them to listen to that night.
  The daily sleep class involve listening to 15 minute audio sessions, which include guided mediation and breathing exercises. Participants will be encouraged to complete classes every day but will be asked to complete classes at least 3 times per week in order to be considered as adhering to the intervention. Participation will be tracked based on participants self-reports in the daily sleep logs. Participants who did not adhere to the intervention will be excluded from per-protocol analyses.
  Participants will complete surveys online at baseline, after 3 weeks, and after 6 weeks. The baseline questionnaires will include demographic information.
  Interventions: Behavioral: Chorus Sleep
- Waitlist (No Intervention): Participants will be placed on a 6 week waitlist to access the chorus sleep app. There will be no daily activities for them to complete during those 6 weeks.
  Participants will complete surveys online at baseline, after 3 weeks, and after 6 weeks. The baseline questionnaires will include demographic information.

INTERVENTIONS:
Behavioral: Chorus Sleep — During the 6-week intervention, participants will receive daily reminders to complete their daily sleep log and a link to a chorus sleep class for them to listen to that night.
  The daily sleep class involve listening to 15 minute audio sessions, which include guided mediation and breathing exercises.
  Arms: Chorus Sleep

SUMMARY:
This pilot study will evaluate the feasibility of a 6-week intervention using Chorus Sleep's ios app to improve sleep quality, reduce stress, and reduce depression and anxiety using a randomized controlled design.

DETAILED DESCRIPTION:
Chorus Sleep is a successful wellness company with a loyal and growing clientele, and considerable qualitative and anecdotal evidence for its efficacy at reducing stress, and improving sleep quality. It builds upon existing meditation and mindfulness practices with well documented efficacy for reducing pain, improving mental health, and reducing stress. Further its innovative approach - including the use of popular music and breathwork patterns that elicit stimulating and novel sensations and physiological activity - may removes barriers to participation and engagement of many traditional meditation and mindfulness practices. Prior research evaluating the efficacy of audio meditation using the Calm app found use of the app for eight weeks significantly decreased daytime fatigue and sleepiness and pre-sleep arousal compared to a wait-list control group. Further, use of the calm app for 8 weeks was associated with greater improvements in depression and anxiety symptoms, and those effects were mediated by lower pre-sleep arousal. This study will investigate whether Chorus Sleep's innovation in auditory app-based sleep inventions will demonstrate similar efficacy.

This study has the following objectives:

1. Pilot a randomized controlled trial on Chorus sleep to evaluate feasibility.
2. Evaluate the effect of Chorus sleep practice at improving sleep quality.
3. Evaluate the effect of Chorus sleep practice at reducing perceived stress, depression, and anxiety, both directly and indirectly through improved sleep quality.
4. Characterize habit formation of Chorus sleep practice

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Have an Apple Iphone 8 or later
* Have a bed to sleep in consistently every night

Exclusion Criteria:

* Narcolepsy
* night shift or shift work for more than 2 nights per week.
* Used the Chorus sleep app more than one time prior to the beginning of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Preliminary effects of the Chorus Sleep app on sleep related impairment, as assessed by changes in participants' self-reported sleep related impairment from pre- to post- 6-week intervention period | Within 24 hours pre-and within 1 week post- 6 week intervention
  Change in total score on the PROMIS Sleep Related Impairment Scale from baseline to 6-week follow-up. Mean scores across the 8 items will be used. Items are a 5-point scale from 1-5. Therefore, the range of possible change scores is from -4 to 4, where a lower negative score corresponds with greater decreases in sleep disturbance, a higher score corresponds with greater increases in sleep disturbance, and 0 indicates no change.

SECONDARY OUTCOMES:
Change in perceived stress | Within 24 hours pre-and within 1 week post- 6 week intervention
  Change in perceived stress on the Perceived Stress Scale-10 from baseline to 6-week follow-up. Mean scores across the 10 items will be used. Items are on a 5-point scale from 1-5. Therefore, the range of possible change scores is from -4 to 4, where lower negative scores correspond with greater decreases in perceived stress, higher positive scores correspond with greater increases in perceived stress, and 0 indicates no change.
Change in depression symptoms | Within 24 hours pre-and within 1 week post- 6 week intervention
  Change in depression symptoms on the PROMIS® Item Bank v1.0 - Emotional Distress - Depression-Short Form 8a from baseline to 6-week follow-up. Mean scores across the 8 items will be used. Items are on a 5-point scale from 1-5. Therefore, the range of possible change scores is from -4 to 4, where lower negative scores correspond with greater decreases in depression, higher positive scores correspond with greater increases in depression, and 0 indicates no change.
Change in anxiety symptoms from baseline to 6-week follow-up. | Within 24 hours pre-and within 1 week post- 6 week intervention
  Change in anxiety symptoms on the PROMIS® Item Bank v1.0 - Emotional Distress - Anxiety - Short Form 8a from baseline to 6-week follow-up. Mean scores across the 8 items will be used. Items are on a 5-point scale from 1-5. Therefore, the range of possible change scores is from -4 to 4, where lower negative scores correspond with greater decreases in anxiety, higher positive scores correspond with greater increases in anxiety, and 0 indicates no change.
Demand, based on frequency of use of the Chorus Sleep app | Recorded continuously throughout 6-week intervention
  The percentage of days in which participants use the chorus sleep app over the course of the 6 week study period.

OTHER OUTCOMES:
Daily self-reported sleep disturbance, as measured by time to fall asleep, on the in-app sleep survey. | Recorded daily throughout the 6 week intervention (intervention group only)
  Daily reports of time to fall asleep reported on the in-app daily sleep survey with options: Fell asleep within 15 minutes, Fell asleep within 16-30 minutes, Fell asleep within 31-60 minutes, Fell asleep after 60 minutes.
Daily self-reported sleep disturbance, as measured by number of awakenings on the in-app sleep survey | Recorded daily throughout the 6 week intervention (intervention group only)
  Daily reports of number of awakenings on the in-app sleep survey with options from 0-more than 4 times in increments of 1.
Daily self-reported sleep disturbance, as measured by total time awake on the in-app sleep survey. | Recorded daily throughout the 6 week intervention (intervention group only)
  Daily reports of number of awakenings on the in-app sleep survey with the following options: 0-30 minutes, 31-60 minutes, 1-2 hours, 2 or more hours
Habit formation | within 1 week post- 6 week intervention
  Habit formation for using the Chorus Sleep App will be measured using an adaptation of the Self-Report Behavioral Automaticity Index. Mean scores will be used across 4 items. Possible scores range from 1-5, where higher scores indicate greater automaticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Online, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made public in an online repository upon publication of results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Study protocol and analytic code will be shared publicly upon publication in a journal and/or upload of to a preprint server.
Access Criteria: Unrestricted